CLINICAL TRIAL: NCT02234583
Title: An Open-label Extension Study of DS-5565 for 52 Weeks in Pain Associated With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS5565-A-E312; 2013-005164-26 (EudraCT Number)
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Pain Associated With Fibromyalgia
Keywords: pain; fibromyalgia
MeSH Terms: conditions — Pain; Fibromyalgia | interventions — mirogabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DS-5565 (Experimental): Participants receive 15 mg DS-5565 administered once or twice daily. Each participant's dose can be titrated up or down based on the investigator's decision. Analysis will be based on the dose modality at the time of data collection.
  Interventions: Drug: DS-5565

INTERVENTIONS:
Drug: DS-5565 — DS-5565 15 mg tablet for oral administration
  Other Names: Investigational product

SUMMARY:
This is an open-label study of DS-5565 in subjects who either completed participation in a preceding Phase 3 study of DS-5565 in fibromyalgia (FM); i.e. DS5565-A-E309 (NCT02146430), DS5565-A-E310 (NCT02187471), or DS5565-A-E311 (NCT02187159) or are de novo subjects. Eligible subjects will be assigned to receive open-label DS-5565 for 52 weeks. All subjects will receive DS-5565 15 mg once daily (QD) for the first three weeks of the treatment period. After three weeks, subjects may be titrated to 15 mg twice daily (BID) based on protocol-specified criteria.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent
* Completed participation (i.e. completed the End-of-Tapering visit) in a preceding study of DS 5565 in FM (DS5565-A-E309, DS5565-A-E310, or DS5565-A-E311)
* Women of child-bearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy during the study and for 4 weeks after study completion
* Able to complete subject-reported questionaires per the investigator's judgement
* The subject must not have experienced any significant safety issues during the preceding study that, in the investigator's judgment, would adversely impact the subject's well-being in the long-term extension

De Novo Subjects

* Age ≥ 18 years
* Able to give written informed consent
* Able to complete subject-reported questionnaires per the investigator's judgment
* At screening, subjects must meet the 1990 American College of Rheumatology (ACR) criteria for FM, i.e. widespread pain present for at least 3 months and pain in at least 11 of 18 specific tender point sites. In addition, the 2010 ACR criteria must be met:

  * Widespread pain index (WPI) ≥ 7 and symptom severity (SS) scale score ≥ 5, or WPI 3 to 6 and SS scale score ≥ 9
  * Symptoms have been present at a similar level for at least 3 months
  * The subject does not have a disorder that would otherwise explain the pain
* ADPS of ≥ 4 on the 11-point numeric rating scale (NRS) over the past 7 days prior to first dose (based on completion of at least 4 daily pain diaries during the 7-day baseline period)
* Subject must have documented evidence of a fundoscopic examination (with pupil dilation) within 12 months prior to screening or at screening
* Women of child-bearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy during the study and for 4 weeks after study completion

Exclusion Criteria:

* Clinically significant unstable neurologic, psychiatric, ophthalmologic, hepatobiliary, respiratory, or hematologic illness or unstable cardiovascular disease (e.g. severe hypotension, uncontrolled cardiac arrhythmia, or myocardial infarction) or any other concurrent disease during the preceding study (for rollover subjects) or within 12 months prior to screening (for de novo subjects) that in the opinion of the investigator would interfere with study participation or assessment of safety and tolerability
* Subjects who are at risk of suicide as defined by their responses to the C-SSRS or in the opinion of the investigator.
* Subjects with severe or uncontrolled depression that, in the judgment of the investigator, makes the subject inappropriate for entry into the study
* Subjects with pain due to other conditions (e.g. DPNP or post-herpetic neuralgia) that, in the opinion of the investigator, would confound assessment or self-evaluation of the pain associated with FM
* Subjects with pain due to any widespread inflammatory musculoskeletal disorder (e.g. rheumatoid arthritis, lupus) or widespread rheumatic disease other than FM.
* Abuse or dependence of prescription medications, street drugs, or alcohol within the last 1 year
* A diagnosis of untreated sleep apnea or initiation of treatment for sleep apnea within the past 3 months
* Known hypersensitivity to α2δ ligands or other components of the study medications
* Pregnancy or breast-feeding, or intent to become pregnant during the study period
* Abnormal investigative tests (i.e. ECGs) and laboratory values judged by the investigator to be clinically significant at the End-of-Treatment visit (Visit - Week 13) in the preceding study (for rollover subjects) or at screening (for de novo subjects), with particular focus on:

For De Novo Subjects Only

* Unable to undergo pre-study washout of prohibited concomitant medications (as listed in Section 5.2.1 of the protocol)
* Current severe or uncontrolled major depressive disorder or anxiety disorders as assessed by the Mini-international Neuropsychiatric Interview (MINI) interview (Version 6.0) at screening are excluded, but mild to moderate major depression or anxiety disorders are permitted provided that the investigator assesses the patient as clinically stable and appropriate for entry into the study
* Any diagnosis of lifetime bipolar disorder or psychotic disorder
* Subject is currently enrolled in or has not yet completed at least 30 days since ending another investigational device or drug study or is receiving other investigational agents
* Subject is an employee of the study center, an immediate family member* of an employee of the study center, or an employee of Daiichi Sankyo, INC Research, or any of the study vendors supporting this study. *(spouse, parent, child, or sibling, whether biological or legally adopted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2485 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (269):
- United States (114):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Anaheim, California
  - Fresno, California
  - Los Alamitos, California
  - Los Angeles, California
  - Newport Beach, California
  - Rancho Mirage, California
  - Roseville, California
  - San Diego, California
  - Santa Ana, California
  - Santa Barbara, California
  - Santa Monica, California
  - Spring Valley, California
  - Thousand Oaks, California
  - Tustin, California
  - Walnut Creek, California
  - Cromwell, Connecticut
  - Bradenton, Florida
  - Brandon, Florida
  - Brooksville, Florida
  - Clearwater, Florida
  - Coral Springs, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Lakeland, Florida
  - Leesburg, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Royal Palm Beach, Florida
  - St. Petersburg, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - Alpharetta, Georgia
  - Atlanta, Georgia
  - Columbus, Georgia
  - Savannah, Georgia
  - Smyrna, Georgia
  - Bolingbrook, Illinois
  - Chicago, Illinois
  - Gurnee, Illinois
  - Melrose Park, Illinois
  - Oak Brook, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - West Des Moines, Iowa
  - Newton, Kansas
  - Shawnee Mission, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Paducah, Kentucky
  - Lake Charles, Louisiana
  - Boston, Massachusetts
  - Fall River, Massachusetts
  - New Bedford, Massachusetts
  - Watertown, Massachusetts
  - Biloxi, Mississippi
  - Hazelwood, Missouri
  - Kansas City, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Blackwood, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Manhasset, New York
  - New York, New York
  - North Massapequa, New York
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Kettering, Ohio
  - Tiffin, Ohio
  - Willoughby, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - Salem, Oregon
  - Tipton, Pennsylvania
  - Wyomissing, Pennsylvania
  - Anderson, South Carolina
  - Fountain Inn, South Carolina
  - Greer, South Carolina
  - Dakota Dunes, South Dakota
  - Rapid City, South Dakota
  - Knoxville, Tennessee
  - New Tazewell, Tennessee
  - Tullahoma, Tennessee
  - Dallas, Texas
  - Lubbock, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Virginia Beach, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Wenatchee, Washington
- Australia (11):
  - Camperdown, New South Wales
  - Campsie, New South Wales
  - Coffs Harbour, New South Wales
  - St Leonards, New South Wales
  - Maroochydore, Queensland
  - Sherwood, Queensland
  - Southport, Queensland
  - Woodville, South Australia
  - Hobart, Tasmania
  - Clayton, Victoria
  - Malvern East, Victoria
- Austria (3):
  - Klagenfurt
  - Senftenberg
  - Vienna
- Bulgaria (8):
  - Burgas
  - Pleven
  - Plovdiv
  - Rousse
  - Sevlievo
  - Sofia
  - Targovishte
  - Varna
- Canada (15):
  - Penticton, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Burlington, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Markham, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
- Chile (2):
  - Antofagasta, Region 11
  - Puerto Varas, Region X
- Czechia (5):
  - Choceň
  - Pilsen
  - Prague
  - Rychnov nad Kněžnou
  - Říčany
- Denmark (2):
  - Aalborg
  - Odense
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (2):
  - Hyvinkää
  - Kuopio
- France (3):
  - Saint-Etienne, Cedex
  - Douai, Nord
  - Élancourt
- Germany (8):
  - Berlin
  - Böhlen
  - Dresden
  - Hanover
  - Leipzig
  - Magdeburg
  - Mainz
  - Stadtroda
- Hungary (4):
  - Balassagyarmat
  - Budapest
  - Debrecen
  - Nyíregyháza
- Latvia (7):
  - Baldone
  - Balvi
  - Jēkabpils
  - Liepāja
  - Ogre
  - Riga
  - Ventspils
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- New Zealand (5):
  - Auckland
  - Hamilton
  - Nelson
  - Tauranga
  - Wellington
- Norway (6):
  - Ålesund
  - Hamar
  - Hønefoss
  - Kløfta
  - Lillehammer
  - Stavanger
- Poland (11):
  - Elblag
  - Gdansk
  - Katowice
  - Krakow
  - Lublin
  - Nadarzyn
  - Nowa Sól
  - Torun
  - Tychy
  - Warsaw
  - Wroclaw
- Portugal (4):
  - Aveiro
  - Guimarães
  - Porto
  - Vila Nova de Gaia
- Puerto Rico (2):
  - Ponce
  - San Juan
- Romania (3):
  - Bacau
  - Bucharest
  - Târgu Mureş
- Russia (4):
  - Krasnoyarsk
  - Moscow
  - Nizhniy Novgarad
  - Stavropol
- Belgrade, Serbia
- Slovakia (7):
  - Banská Bystrica
  - Bratislava
  - Dubnica nad Váhom
  - Galanta
  - Krompachy
  - Piešťany
  - Prešov
- Slovenia (2):
  - Ljubljana
  - Slovenj Gradec
- South Africa (7):
  - Bayview, Chatsworth
  - Johannesburg, Gautang
  - Pretoria, Gautang
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
  - Somerset West, Western Cape
  - Stellenbosch
- Spain (4):
  - Santiago de Compostela, A Coruna
  - Barcelona
  - Granada
  - Madrid
- Ukraine (8):
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kherson
  - Kyiv
  - Lviv
  - Vinnytsia
  - Zaporizhzhia
- United Kingdom (16):
  - Penzance, Cornwall
  - Chesterfield, Derbyshire
  - Romford, Essex
  - Manchester, Greater Manchester
  - Blackpool, Lancashire
  - Thornton-Cleveleys, Lancashire
  - Wigan, Lancashire
  - Stourton, Leeds
  - Salford, Manchester
  - Southport, Merseyside
  - Wellingborough, Northamptonshire
  - Belfast, Northern Ireland
  - Cannock, Staffordshire
  - North Shields, Tyne and Wear
  - Atherstone, Warwickshire
  - Torpoint

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Arnold LM, Whitaker S, Hsu C, Jacobs D, Merante D. Efficacy and safety of mirogabalin for the treatment of fibromyalgia: results from three 13-week randomized, double-blind, placebo- and active-controlled, parallel-group studies and a 52-week open-label extension study. Curr Med Res Opin. 2019 Oct;35(10):1825-1835. doi: 10.1080/03007995.2019.1629757. Epub 2019 Jul 9. PMID 31284771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2485 participants who met all inclusion and no exclusion criteria enrolled from 04 Feb 2015 to 19 Apr 2017 at 406 clinic sites. Of the 2485 enrolled, 397 discontinued prior to randomization. A total of 2088 participants received study treatment.
Pre-assignment Details: Participants who completed the double-blind studies of DS-5565 in fibromyalgia were eligible to Rollover to this open-label extension study (referred to as Rollover participants). Participants who did not participate in a preceding double-blind study (referred to as De Novo participants) could be enrolled at the discretion of the Sponsor.
Groups:
- DS-5565 15 mg QD Modal: Participants received DS-5565 in a preceding Phase 3 study of DS-5565 in fibromyalgia (DS5565-A-E309 [NCT02146430], DS5565-A-E310 [NCT02187471], or DS5565-A-E311 [NCT02187159]) and received 15 mg DS-5565 administered once daily (QD) for the first 3 weeks. After 3 weeks, participants could be titrated to BID. This group includes both rollover and De Novo QD modal.
- DS-5565 15 mg BID Modal: Participants received DS-5565 in a preceding Phase 3 study of DS-5565 in fibromyalgia (DS5565-A-E309 [NCT02146430], DS5565-A-E310 [NCT02187471], or DS5565-A-E311 [NCT02187159]) and received 15 mg DS-5565 administered once daily (QD) for the first 3 weeks. After 3 weeks, participants could be titrated to BID. This group includes both rollover and De Novo twice daily (BID) modal.
Period: Overall Study
Arm/Group | DS-5565 15 mg QD Modal | DS-5565 15 mg BID Modal
Started | 847 | 1241
Completed | 434 | 685
Not Completed | 413 | 556
Not completed — Adverse Event | 172 | 156
Not completed — Withdrawal by Subject | 109 | 157
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 58 | 103
Not completed — Protocol Violation | 35 | 42
Not completed — Other | 39 | 97

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics are derived from the Safety Analysis Set.
Groups:
- DS-5565 15 mg BID Modal: Participants received DS-5565 in a preceding Phase 3 study of DS-5565 in fibromyalgia (DS5565-A-E309 [NCT02146430], DS5565-A-E310 [NCT02187471], or DS5565-A-E311 [NCT02187159]) and received 15 mg DS-5565 administered once daily (QD) for the first 3 weeks. After 3 weeks, participants could be titrated to twice daily (BID). This group includes both rollover and De Novo BID modal.
- Total: Total of all reporting groups
Arm/Group | DS-5565 15 mg QD Modal | DS-5565 15 mg BID Modal | Total
Number analyzed (Participants) | 847 | 1241 | 2088
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 750 | 1128 | 1878
  >=65 years | 97 | 113 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (11.18) | 49.3 (11.94) | 50.2 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 770 | 1130 | 1900
  Male | 77 | 111 | 188
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 82 | 113 | 195
  White | 740 | 1101 | 1841
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 18 | 37
Region of Enrollment [Number; unit: participants]
  United States | 569 | 913 | 1879
  Czechia | 11 | 27 | 38
  Portugal | 0 | 4 | 4
  Russia | 10 | 1 | 11
  Austria | 5 | 10 | 15
  Latvia | 11 | 8 | 19
  Poland | 16 | 24 | 40
  Slovakia | 14 | 4 | 18
  Slovenia | 4 | 3 | 7
  Bulgaria | 14 | 6 | 20
  Chile | 1 | 4 | 5
  France | 4 | 2 | 6
  Lithuania | 3 | 1 | 4
  Serbia | 0 | 3 | 3
  Romania | 3 | 1 | 4
  Hungary | 6 | 1 | 7
  Ukraine | 73 | 59 | 264
  United Kingdom | 14 | 27 | 41
  Spain | 8 | 19 | 27
  New Zealand | 7 | 11 | 18
  Canada | 17 | 35 | 52
  Norway | 12 | 30 | 42
  Finland | 0 | 1 | 1
  Denmark | 7 | 5 | 12
  South Africa | 9 | 10 | 38
  Australia | 5 | 8 | 13
  Germany | 22 | 16 | 38
  Estonia | 2 | 8 | 10

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Pain Score (ADPS) for DS-5565
Description: Average of daily pain scores are reported by the participant and best describes his or her worst pain over the previous 24 hours. A daily pain score has a scale of 0 = no pain to 10 = worst possible pain.
Time Frame: Day 0 (baseline) up to to Week 52 postdose
Population: Average daily pain score was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Rollover DS-5565 15 mg QD Modal; Rollover DS-5565 15 mg BID Modal: Participants received DS-5565 in a preceding Phase 3 study of DS-5565 in fibromyalgia (DS5565-A-E309 [NCT02146430], DS5565-A-E310 [NCT02187471], or DS5565-A-E311 [NCT02187159]) and received 15 mg DS-5565 administered once daily (QD) for the first 3 weeks. After 3 weeks, participants could be titrated to twice daily (BID). Participants were reported by their modal dose or dose received most frequently.
- De Novo DS-5565 15 mg QD Modal; De Novo DS-5565 15 mg BID Modal: Participants with no prior exposure to DS-5565 and received 15 mg DS-5565 administered once daily (QD) for the first 3 weeks. After 3 weeks, participants could be titrated to twice daily (BID). Participants were reported by their modal dose or dose received most frequently.
Arm/Group | Rollover DS-5565 15 mg QD Modal | Rollover DS-5565 15 mg BID Modal | De Novo DS-5565 15 mg QD Modal | De Novo DS-5565 15 mg BID Modal
Number analyzed (Participants) | 578 | 962 | 269 | 279
score on a scale
  Baseline: number analyzed (Participants) | 562 | 940 | 264 | 274
  Baseline | 4.77 (2.23) | 5.58 (2.22) | 7.08 (1.40) | 7.38 (1.37)
  Week 13: number analyzed (Participants) | 398 | 809 | 165 | 237
  Week 13 | 3.47 (2.11) | 4.36 (2.32) | 3.21 (2.20) | 4.06 (2.37)
  Week 24: number analyzed (Participants) | 340 | 661 | 148 | 194
  Week 24 | 3.28 (2.08) | 4.24 (2.35) | 3.0 (2.14) | 4.0 (2.38)
  Week 36: number analyzed (Participants) | 301 | 552 | 126 | 156
  Week 36 | 3.20 (2.06) | 4.25 (2.34) | 2.74 (2.23) | 3.95 (2.59)
  Week 48: number analyzed (Participants) | 269 | 470 | 121 | 137
  Week 48 | 3.22 (2.16) | 4.25 (2.37) | 2.46 (2.15) | 3.80 (2.61)
  Week 52: number analyzed (Participants) | 245 | 432 | 109 | 121
  Week 52 | 3.20 (2.18) | 4.26 (2.42) | 2.31 (1.94) | 3.80 (2.70)

2. Secondary Outcome: Number of Participants With Much Improved or Better (≤2) Status in Status at Week 52 As Assessed by the Patient-Rated Global Impression of Change
Description: Patient-rated global impression of change (PGIC) on a categorical scale from 1 = very much improved to 7 = very much worse. The number of participants with "much improved or better" status are reported.
Time Frame: Week 52 postdose
Population: Patient Global Impression of Change was assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Rollover DS-5565 15 mg QD Modal | Rollover DS-5565 15 mg BID Modal | De Novo DS-5565 15 mg QD Modal | De Novo DS-5565 15 mg BID Modal
Number analyzed (Participants) | 578 | 962 | 269 | 279
Participants | 208 | 333 | 96 | 92

3. Secondary Outcome: Hospital Anxiety Depression Scale (HADS) Depression and Anxiety Scores for DS-5565
Description: The HADS questionnaire is a self-assessment scale to assess symptoms of anxiety and depression. The instrument consists of 7 questions related to anxiety and 7 related to depression, each rated on a 4-point scale from 0 to 3, where higher scores indicate greater anxiety or depression. Scores for anxiety and depression are independently summed to compute HADS-Anxiety and HADS-Depression subscale scores, with ranges from 0 to 21, where higher scores indicate greater severity.
Time Frame: Day 0 (baseline) up to Week 52 postdose
Population: HADS-Depression and Anxiety was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Rollover DS-5565 15 mg QD Modal; Rollover DS-5565 15 mg BID Modal: Participants received DS-5565 in a preceding Phase 3 study of DS-5565 in fibromyalgia (DS5565-A-E309 [NCT02146430], DS5565-A-E310 [NCT02187471], or DS5565-A-E311 [NCT02187159]) and received 15 mg DS-5565 administered once daily (QD) for the first 3 weeks. After 3 weeks, participants could be titrated to twice daily (BID). Participants were reported by their modal dose or dose received most frequently.
  DS-5565: DS-5565 15 mg tablet for oral administration
- De Novo DS-5565 15 mg QD Modal; De Novo DS-5565 15 mg QID Modal: Participants with no prior exposure to DS-5565 and received 15 mg DS-5565 administered once daily (QD) for the first 3 weeks. After 3 weeks, participants could be titrated to twice daily (BID). Participants were reported by their modal dose or dose received most frequently.
  DS-5565: DS-5565 15 mg tablet for oral administration
Arm/Group | Rollover DS-5565 15 mg QD Modal | Rollover DS-5565 15 mg BID Modal | De Novo DS-5565 15 mg QD Modal | De Novo DS-5565 15 mg QID Modal
Number analyzed (Participants) | 578 | 962 | 269 | 279
score on a scale
  Anxiety Subscale Baseline: number analyzed (Participants) | 520 | 894 | 266 | 271
  Anxiety Subscale Baseline | 5.7 (3.86) | 7.2 (4.05) | 6.9 (3.97) | 7.4 (4.21)
  Anxiety Subscale Week 52: number analyzed (Participants) | 308 | 539 | 124 | 142
  Anxiety Subscale Week 52 | 4.8 (3.71) | 7.0 (4.03) | 4.4 (3.29) | 5.7 (3.88)
  Depression Subscale Baseline: number analyzed (Participants) | 520 | 894 | 266 | 271
  Depression Subscale Baseline | 5.1 (4.18) | 6.3 (4.34) | 5.6 (4.06) | 5.7 (4.10)
  Depression Subscale Week 52: number analyzed (Participants) | 308 | 539 | 124 | 142
  Depression Subscale Week 52 | 3.5 (3.47) | 4.8 (4.01) | 2.8 (3.11) | 3.9 (4.00)

4. Secondary Outcome: EuroQol Five Dimensions Questionnaire (EQ-5D) Measure for DS-5565
Description: The EQ-5D is an instrument that shows high construct validity and responsiveness in patients with chronic pain and has been used specifically in fibromyalgia. The EQ-5D includes a descriptive section with 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that are combined into an overall health utilities index, and an NRS (100 mm VAS) that measures perception of overall health, with 0 indicating worst health and 100 representing best imaginable health.
Time Frame: Day 0 (baseline) up to Week 52 postdose
Population: EQ-5D was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover DS-5565 15 mg QD Modal | Rollover DS-5565 15 mg BID Modal | De Novo DS-5565 15 mg QD Modal | De Novo DS-5565 15 mg BID Modal
Number analyzed (Participants) | 578 | 962 | 269 | 279
units on a scale
  Total Score Baseline: number analyzed (Participants) | 520 | 894 | 266 | 271
  Total Score Baseline | 0.70 (0.17) | 0.64 (0.19) | 0.62 (0.16) | 0.61 (0.18)
  Total Score Week 52: number analyzed (Participants) | 308 | 539 | 124 | 142
  Total Score Week 52 | 0.76 (0.16) | 0.70 (0.20) | 0.81 (0.15) | 0.77 (0.17)

5. Secondary Outcome: Short Form-36 (SF-36) Measure for DS-5565
Description: The SF-36 is a 36-question health survey that measures functional health and well-being from the participant's point of view. It is a measure of physical and mental health used across various disease areas, including fibromyalgia. The SF-36 physical component summary and mental component summary scales range from 0 to 100 where lower scores indicate more disability (worse health) and higher scores represent less disability (better health). The physical component summary (PCS) and mental component summary (MCS) total scores at baseline and Week 52 are reported.
Time Frame: Day 0 (baseline) to Week 52 postdose
Population: SF-36 was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rollover DS-5565 15 mg QD Modal | Rollover DS-5565 15 mg BID Modal | De Novo DS-5565 15 mg QD Modal | De Novo DS-5565 15 mg BID Modal
Number analyzed (Participants) | 578 | 962 | 269 | 279
score on a scale
  Physical Component Summary Baseline: number analyzed (Participants) | 520 | 894 | 266 | 270
  Physical Component Summary Baseline | 37.91 (8.86) | 35.13 (8.55) | 34.41 (8.58) | 32.12 (7.85)
  Physical Component Summary Week 52: number analyzed (Participants) | 308 | 539 | 124 | 142
  Physical Component Summary Week 52 | 42.96 (8.52) | 39.09 (9.38) | 45.61 (9.63) | 42.31 (10.47)
  Mental Component Summary Baseline: number analyzed (Participants) | 520 | 894 | 266 | 270
  Mental Component Summary Baseline | 50.12 (10.19) | 47.76 (11.15) | 47.54 (10.98) | 47.92 (11.46)
  Mental Component Summary Week 52: number analyzed (Participants) | 308 | 539 | 124 | 142
  Mental Component Summary Week 52 | 52.63 (9.61) | 49.15 (11.24) | 52.75 (8.02) | 50.49 (10.54)

6. Secondary Outcome: Pain-Associated Sleep Interference as Assessed by Average Daily Sleep Interference Score (ADSIS) for DS-5565
Description: Pain-associated sleep interference was assessed using electronic daily diaries using an 11-point numeric rating scale (NRS) for pain, ranging from 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep, unable to sleep). ADSIS is the mean value of all available recordings of the respective week. For rollover participants, the baseline scores from the End-of-Tapering period in the preceding study are reported. For de novo participants, the baseline scores are derived from the 7 days prior to the start of treatment.
Time Frame: Day 0 (baseline) up to Week 52 postdose
Population: Average Daily Sleep Interference Score was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rollover DS-5565 15 mg QD Modal | Rollover DS-5565 15 mg BID Modal | De Novo DS-5565 15 mg QD Modal | De Novo DS-5565 15 mg BID Modal
Number analyzed (Participants) | 578 | 962 | 269 | 279
score on a scale
  Baseline: number analyzed (Participants) | 562 | 940 | 264 | 274
  Baseline | 3.84 (2.41) | 4.74 (2.52) | 6.71 (1.70) | 6.82 (1.82)
  Week 13: number analyzed (Participants) | 398 | 809 | 165 | 237
  Week 13 | 2.56 (2.16) | 3.18 (2.50) | 2.50 (2.15) | 3.13 (2.51)
  Week 24: number analyzed (Participants) | 340 | 661 | 148 | 194
  Week 24 | 2.34 (1.96) | 3.09 (2.50) | 2.36 (2.18) | 3.19 (2.48)
  Week 36: number analyzed (Participants) | 301 | 552 | 126 | 156
  Week 36 | 2.25 (1.98) | 3.09 (2.50) | 2.19 (2.20) | 3.11 (2.63)
  Week 48: number analyzed (Participants) | 269 | 470 | 121 | 137
  Week 48 | 2.32 (2.07) | 3.22 (2.56) | 1.87 (2.05) | 3.02 (2.64)
  Week 52: number analyzed (Participants) | 245 | 432 | 109 | 121
  Week 52 | 2.22 (2.06) | 3.19 (2.63) | 1.79 (1.86) | 3.09 (2.71)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to 4 weeks after last dose, up to 2 years 3 months.
Description: A TEAE was any adverse event that emerged on or after the first dosing of open-label extension (OLE) medication and during study treatment up to 4 weeks after the last dose of OLE medication (having been absent prior to treatment) or worsened relative to the pre-OLE treatment state.
Groups:
- DS-5565 15 mg QD Modal: Participants received DS-5565 in a preceding Phase 3 study of DS-5565 in fibromyalgia (DS5565-A-E309, DS5565-A-E310, or DS5565-A-E311) and received 15 mg DS-5565 administered once daily (QD) for the first 3 weeks. After 3 weeks, participants could be titrated to BID. This group includes both rollover and De Novo QD modal.
- DS-5565 15 mg BID Modal: Participants received DS-5565 in a preceding Phase 3 study of DS-5565 in fibromyalgia (DS5565-A-E309, DS5565-A-E310, or DS5565-A-E311) and received 15 mg DS-5565 administered once daily (QD) for the first 3 weeks. After 3 weeks, participants could be titrated to BID. This group includes both rollover and De Novo twice daily (BID) modal.
Arm/Group | DS-5565 15 mg QD Modal | DS-5565 15 mg BID Modal
All-Cause Mortality (participants affected / at risk) | 3/847 | 2/1241
Serious Adverse Events (participants affected / at risk) | 41/847 | 94/1241
Other Adverse Events (participants affected / at risk) | 669/847 | 1056/1241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-5565 15 mg QD Modal (N=847) | DS-5565 15 mg BID Modal (N=1241)
Appendicitis (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Convulsion (Nervous system disorders) | 0 | 3
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 4
Oedema peripheral (General disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Suicidal ideation (Psychiatric disorders) | 3 | 3
Suicide attempt (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Hepatic enzyme increased (Investigations) | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 1
Abscess limb (Infections and infestations) | 0 | 1
Chronic hepatitis C (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Infectious colitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Meningitis aseptic (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerous fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine phosphokinase abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Spine malformation (Congenital, familial and genetic disorders) | 0 | 1
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Bereavement (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DS-5565 15 mg QD Modal (N=847) | DS-5565 15 mg BID Modal (N=1241)
Upper respiratory tract infection (Infections and infestations) | 43 | 134
Urinary tract infection (Infections and infestations) | 51 | 107
Nasopharyngitis (Infections and infestations) | 47 | 110
Sinusitis (Infections and infestations) | 36 | 89
Dizziness (Nervous system disorders) | 134 | 148
Headache (Nervous system disorders) | 123 | 158
Somnolence (Nervous system disorders) | 130 | 102
Drug withdrawal syndrome (General disorders) | 61 | 135
Fatigue (General disorders) | 76 | 83
Oedema peripheral (General disorders) | 52 | 82
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 89
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 88
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 64
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 26 | 62
Nausea (Gastrointestinal disorders) | 61 | 113
Diarrhoea (Gastrointestinal disorders) | 40 | 97
Weight increased (Investigations) | 83 | 207
Insomnia (Psychiatric disorders) | 34 | 63
Vision blurred (Eye disorders) | 26 | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT02234583/Prot_SAP_000.pdf